CLINICAL TRIAL: NCT06024941
Title: Re-induction of a Systemic Immune Response After Initial Response With Immune Therapy With Single-dose Radiotherapy in Metastatic or Locally Recurrent Lung Cancer: A Prospective Phase II Trial (Re-Induce 2)
Brief Title: Re-induction of a Systemic Immune Response in Metastatic or Locally Recurrent Lung Cancer
Acronym: Re-Induce 2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Submission not finished
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Re-Induce 2
Record Dates: First submitted 2023-08-22; First posted 2023-09-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer Stage IV
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation (Experimental): Radiation to one progressive lesion
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiation to one or more progressive lesions. Preferably 1x10Gy, but also 3x8Gy, 10x 3Gy, 5x4Gy or 1x20-24Gy is possible.

SUMMARY:
Patients with metastatic non-small cell lung cancer (NSCLC) who after an initial response to immunotherapy of chemo-immunotherapy show diffuse disease progression are treated with chemotherapy, with a median PFS of about 3 months and a high incidence of important toxicity or by continuation of immune therapy when the growth rate of the tumours is low. In a previous study, it was showed that irradiating a single metastatic lesion and continuation of immune therapy resulted in a median PFS time was 4.9 months (95% CI, 3.0-7.0 months). At three months of follow-up, the PFS rate was 62.5%, at six months 37.5% and at 12 months 17.9%. The median OS for all patients was 14.9 months (95% CI, 12.2-21.5 months). Toxicity was hardly observed. This was obtained with a few fractions of radiotherapy. There is biological rationale to deliver this radiation in a single fraction of 10 Gy.

Objective: The primary objective is to investigate if a single fraction of 10 Gy is not inferior to a more fractionated schedule, which would add to the convenience for the patient, even less toxicity and costs.

Study design: Prospective, single-arm phase II trial. Study population: Patients with stage IV NSCLC who initially showed a partial or complete remission under immune therapy alone or concurrent immune therapy and chemotherapy and now show progressive disease according to RECIST 1.1 criteria. At least two different lesions should show progressive disease. Patients should be able to continue the same immune therapy (i.e. no adverse events grade 3 or more).

Intervention: Patients continue the same immune therapy they already received and get radiotherapy to one progressing lesion. The lesion may or may not be symptomatic. The preferred radiotherapy dose is 10 Gy in 1 fraction, but other fractionation schedules (e.g. 24 Gy/ 3 fractions, 30 Gy/ 10 fractions, 20 Gy/ 5 fractions, 20-24 Gy / 1 fraction for stereotactic radiotherapy for brain metastases), including so-called isotoxic strategies are allowed if these are standard for a certain location or palliative indication in the body.

Main study parameters/endpoints: Progression-free survival (PFS).

DETAILED DESCRIPTION:
Metastatic non-small cell lung cancer (NSCLC) has always had a remarkably high mortality, with a 5-year overall survival (OS) rate of only 6%.However, immune checkpoint inhibitors (ICI) targeting the programmed death protein (PD-1)/programmed death-ligand 1 (PD-L1) axis have changed this outcome significantly. Patients with NSCLC who have been treated with ICI, either as monotherapy or in combination with chemotherapy, are surviving longer as compared to patients receiving chemotherapy alone,5-14 with 5-year OS rates as high as 15-30%.This has led to the implementation of ICI in clinical practice, namely in patients with metastatic NSCLC without specific gene alterations.

Despite overall improved survival rates, a considerable number of patients fail to achieve a response when treated with ICI (primary resistance) or develop resistance after an initial period of clinical and radiological response (acquired resistance). Resistance to ICI is thought to be the result of tumor cell intrinsic factors and an immunosuppressive tumor microenvironment, resulting in the suppression of effective anti-tumor immunity. Currently, treatment options in case of resistance to PD1/PD-L1 blockade are limited, with chemotherapy being standard of care outside clinical trials. The PFS and OS in fit patients receiving double-agent chemotherapy after progression are approximately 5 and 12 months, while for those receiving single-agent chemotherapy only 4 and 10 months, respectively. Therefore, exploring treatments for overcoming ICI resistance is warranted.

Radiation therapy (RT) is an effective and common treatment in advanced NSCLC, playing a major role in symptom control, improving quality of life and potentially survival in oligometastatic disease. Moderately hypofractionated RT to tumor or metastases, while sparing lymphoid tissues such as lymph nodes, bone marrow and the circulating blood pool, was shown to enhance the immune response with clinical benefit.

Acquired immunotherapy resistance is a common event in NSCLC, with most patients exhibiting progression within the first 6 months (20%) or the first year of treatment (35%). Clinical trials directed at overcoming immunotherapy resistance in NSCLC have mainly focused on the escalation of systemic therapy by dual checkpoint blockade or by addition of supporting substances. A phase II trial investigated the role of durvalumab plus tremelimumab in this setting and showed no benefit. In contrast, the randomized phase II study of ramucirumab and pembrolizumab showed improved OS of 14.5 months versus 11.6 months with standard of care. In other trials investigating chemotherapy plus immunotherapy after ICI-resistance, the continuation of immunotherapy beyond disease progression also resulted in improved outcomes compared to patients receiving chemotherapy alone.

Since previous works have demonstrated that the combination of ICI with RT in immunotherapy-naïve patients has a relevant impact on PFS, OS and rate of abscopal responses, local radiation has also been considered a viable option for overcoming immunotherapy resistance.

In the predecessor of the current study, "Re-induction of a systemic immune response after initial response with immune therapy with radiotherapy in metastatic or locally recurrent lung cancer: A prospective phase II trial", NCT03406468, the clinical benefit of adding radiotherapy to immune therapy was investigated. The results of a similar study at the University Hospital Freiburg, Germany, RadImmun-NSCLC ("Evaluation of systemic effects of combined palliative radiation therapy and immunotherapy in patients with metastatic non-small cell lung cancer after insufficient response to immune checkpoint blockade", DRKS00013531), were pooled [submitted manuscript].

A total of 48 patients were enrolled between March 2018 and September 2021 in Freiburg and Maastricht, 25 patients within the RadImmun-NSCLC trial and 23 patients within the Re-Induction trial. All patients had stage IV NSCLC, with the majority having adenocarcinoma.

Importantly, following progression, 21.9% of patients were salvaged again by using local irradiation.

The median PFS time was 4.9 months (95% CI, 3.0-7.0 months). At three months of follow-up, the PFS rate was 62.5%, at six months 37.5% and at 12 months 17.9%.

With 62.5% of patients having no tumor progression three months after RT, the results of the trials exceeded the initial hypothesis and suggest that radiation can boost the systemic immune response, at least temporarily. Moreover, the median OS following RT was 14.9 months, which is significantly higher than historical data on chemotherapy in the same context. These results are similar to those obtained by escalation of systemic treatment with dual checkpoint blockade or the combination of ramucirumab and pembrolizumab. However, in contrast to the strategy to add another pharmacological agent, the rate of high-grade adverse events was minimized in the study by keeping the immune treatment unchanged (25% versus 34-42%). The results are in line with previous studies showing low toxicity of the combination between stereotactic RT and immunotherapy.

Similar positive results were achieved by a prospective trial investigating the RT-ICI combination in oligo progressive metastatic NSCLC and melanoma patients. As approximately 40% of patients had malignant melanoma and 50% were primarily refractory to ICI, a clear interpretation of the results in the context of acquired resistance in NSCLC is not possible. Furthermore, patients were not classified as progressive in this trial as long as they could be salvaged by further RT, which could explain the unexpectedly high median PFS of 14.2 months.

In a multicenter randomized phase 2 trial evaluating durvalumab plus tremelimumab and RT for NSCLC in the same setting, neither low-dose nor hypofractionated RT could enhance the systemic response compared to the dual checkpoint blockade alone. However, median PFS values were generally higher in this trial (4-4.6 months) as compared to standard chemotherapy. In the study, the initial ICI was maintained, and the addition of RT alone led to comparable PFS values of 4.9 months, with about 18% of patients still having no further progression at 12 months.

There is evidence that particular dose fractionations may lead to a more pronounced immune modulation than others. Taking into consideration the heterogeneous dose regimens in our pooled cohort, it appears that any type of hypofractionated RT might be efficient in prolonging PFS. A recently published study suggests that this beneficial effect might be dependent on tumor aneuploidy, which could be used as a prognostic biomarker. In Maastro's trial, the aggressiveness of the tumor, characterized by its metastasis growth rate, seemed to impact outcome, with slower-growing tumors having an improved PFS. Some studies also found a significant correlation between pretherapeutic tumor growth and OS, however others have not. Following RT, the lesion velocity decreased, attaining at least stable disease in over 90% of patients for a median of 6.2 months.

In Maastro's trial, at least one metastasis had to be left untreated for follow-up. Nevertheless, the incidental partial irradiation of all measurable lesions was noticed in 11 patients, who also showed an improved outcome. The partial irradiation of metastases in combination with immunotherapy has been suggested to have good local efficacy, and the irradiation of all lesions to improve outcome. However, this is only possible in oligometastatic disease. The trial shows that all metastatic NSCLC patients benefit from RT of selected lesions, presumably with improved results in those with a slower tumor dynamic.

Studies in Maastricht and in Freiburg in patients with NSCLC are indicative that the immune activation already occurs within days after a single fraction of radiotherapy, likely after 10 Gy. Therefore, a single dose of radiation might be as effective to stimulate the immune system as a hypofractionated regimen such as 24 Gy/ 3 fractions in our previous study, while improving the convenience of the treatment for patients, decrease the costs of the intervention and even further reduce toxicity. A single fraction of 10 Gy has been extensively investigated and used for palliative radiotherapy and has been shown to be safe.

The aim of the present study is therefore to investigate if a single fraction of 10 Gy will also lead to similar disease control rates in patients showing progressive disease after an initial response of immunotherapy as 3x8 Gy fractionated radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV NSCLC
* An initial partial or complete remission under immune therapy alone or concurrent immune therapy and chemotherapy
* Subsequently progressive disease according to RECIST 1.1 criteria
* Considered by the treating physician to be able to continue the same immune treatment as standard of care
* At least two different lesions should show progressive disease
* At least one progressing lesion should be eligible for radiation

Exclusion Criteria:

* Patients with any grade 3 or higher toxicity from previous therapy
* Patients who are not eligible for continuation of the immune therapy according to standard practice
* Corticosteroids in a dose above 10 mg prednisone or equivalent per day. Corticoids used as supportive therapy for systemic or radiotherapy are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free | 3 months after radiotherapy
  Progression-free survival (PFS)

SECONDARY OUTCOMES:
Regression | 3 months after radiotherapy
  Number of patients who show regression of the irradiated lesion
Remission rate | 3 months after radiotherapy
  Number of patients who show remission (RECIST 1.1) of the non-irradiated lesion(s)
Toxicity | 3 months after radiotherapy
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0Toxicity (CTCAE 4.0) of this combination of remission and regression
Overall survival | 3 months after radiotherapy
  Overall survival (OS)
PFS second course | 3 months after radiotherapy
  PFS of patients who received a second course of radiotherapy at the time of disease progression
Number | 3 months after radiotherapy
  Number of patients who received a second course of radiotherapy at the time of disease progression
Relation between the growth rate of the fastest growing metastasis in the 3 months preceding radiotherapy and PFS | 3 months after radiotherapy
  Relation between the growth rate of the fastest growing metastasis in the 3 months preceding radiotherapy and PFS

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — Maastro
Locations (1):
- Maastricht Radiation Oncology (Maastro), Maastricht, Netherlands